CLINICAL TRIAL: NCT01409083
Title: Evaluating the Use of Intravenous Bicarbonate as a Tool to Verify the Intravascular Position of an IV Catheter in Children
Brief Title: Intravenous Sodium Bicarbonate Verifies Intravenous Position of Catheters in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Dr. Ilan Keidan, director of pediatric anesthesia, Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: SHEBA-11-8207-IK-CTIL
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Verifying the Correct Position of Intravenous Catheters
Keywords: infiltration; extravasation; end-tidal carbon dioxide; sodium bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- intravenous bicarbonate (Experimental): Diluted sodium bicarbonate will be injected to s new IV catheter expecting a rise in end-tidal CO2
  Interventions: Device: intravenous sodium bicarbonate
- control (Placebo Comparator): equal volume of normal saline will be randomely injected
  Interventions: Device: intravenous sodium bicarbonate

INTERVENTIONS:
Device: intravenous sodium bicarbonate — Dilted sodium bicarbonate 2.1%

SUMMARY:
Sodium bicarbonate injected into a blood vessel transforms to carbon dioxide and water. The increase in carbon dioxide production can be detected by measuring the exhaled carbon dioxide in the lungs.

This study is conducted to access the clinical application of measuring exhaled carbon dioxide to verify the correct position of intravenous catheters.Once the catheter is in the correct position the injected bicarbonate will be detected as a distinct elevation of exhaled carbon dioxide. A similar study was already performed in adults and was found useful. The investigators now extend the clinical application to children.

DETAILED DESCRIPTION:
Extravasation is the unintentional injection or leakage of fluids into the perivascular or subcutaneous space resulting in potential tissue injury. This prospective controlled study, will assesse the diagnostic utility of using intravenous diluted sodium bicarbonate to confirm placement of intravenous (IV) catheters in ventilated children. Diluted sodium bicarbonate will be created using undiluted standard 8.4% (1 meq/mL) sodium bicarbonate mixed in a 1:3 ratio with sterile water to achieve a final diluted concentration of 2.1% (0.25 mEq/mL). In 20 ASA I-II mechanically ventilated children age 2-8 years, the effects of 1 ml/kg of diluted 2.1% sodium bicarbonate or 0.9% normal saline,injected in a randomized order, will be analyzed. All children will have venous blood samples taken prior to injection and 10 minutes after injection for analysis of venous blood pH and electrolytes.

ELIGIBILITY:
Inclusion Criteria:

* ASA I,II
* age 2-8 years

Exclusion Criteria:

* ASA III or higher

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
increase in exhaled carbon dioxide | 0.5-10.00 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel